CLINICAL TRIAL: NCT04590547
Title: Safety, Tolerability and Efficacy and Dose Response of GLS-1027 in the Prevention of Severe Pneumonitis Caused by SARS-CoV-2 Infection
Brief Title: GLS-1027 for the Prevention of Severe Pneumonitis Caused by SARS-CoV-2 Infection (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GeneOne Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GLS27-005
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Pneumonitis; SARS-CoV Infection
Keywords: COVID-19
MeSH Terms: conditions — Pneumonia; Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GLS-1027 120 mg (Experimental): One 120 mg pill of GLS-1027 + 2 Placebo pills given by mouth once daily
  Interventions: Drug: GLS-1027
- GLS-1027 360 mg (Experimental): Three 120 mg pills of GLS-1027 given by mouth once daily
  Interventions: Drug: GLS-1027
- Placebo (Placebo Comparator): Three Placebo pills given by mouth once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLS-1027 — GLS-1027 is an oral medication with high bioavailability that has IL-6 and IL-1β inhibitory activity.
  Arms: GLS-1027 120 mg; GLS-1027 360 mg
Drug: Placebo — Placebo looks like GLS-1027
  Arms: Placebo

SUMMARY:
This clinical trial will evaluate the safety, tolerability and efficacy of GLS-1027 in the prevention of severe pneumonitis caused by SARS-CoV-2 infection

DETAILED DESCRIPTION:
This Phase II randomized, double-blind, placebo-controlled, study will assess 2 different doses of GLS-1027 in the prevention of severe pneumonitis among those hospitalized with PCR confirmed SARS-CoV-2 infection. Subjects will be randomized at a 1:1:1 ratio to either Standard of Care (SOC) plus placebo, or SOC plus GLS-1027 at either 120 mg or 360 mg daily. Clinical status will be monitored through 56 days from the initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able to provide consent
* Able and willing to comply with study procedures
* Diagnosis of PCR confirmed SARS-CoV-2
* Enrollment within 72 of hospitalization
* WHO COVID-19 classification level 3 or 4

Exclusion Criteria:

* Pregnant or lactating
* Need for mechanical ventilation, non-invasive ventilation (NIV), or high-flow O2 (≥60%) via face mask
* Calculated GFR < 60 (Cockcroft-Gault)
* Meets treatment algorithm criteria for treatment with a non-study immune modulator
* Pre-study or planned treatment with a non-study immune modulator
* Participation in a COVID-19 clinical trial that includes prescription of a drug with anti-cytokine activity
* Status post transplantation of an organ, bone marrow, or body part
* Treatment within the past 60 days with a chemotherapeutic agent
* Diagnosis of leukemia or lymphoma
* WHO COVID-19 classification level of 5 or greater
* Unable to take oral medication
* Grade 3 or greater laboratory abnormalities as characterized by CTCAE v5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2023-07-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- Baton Rouge General Medical Center, Baton Rouge, Louisiana, United States
- Bulgaria (5):
  - MHAT Kozlodui, Kozloduy
  - SHATPPD d-r Dimitar Gramatikov, Department of Pneumology, Rousse
  - UMHAT MEDICA RUSE LTD, Internal Diseases Department/Covid, Rousse
  - Military MHAT Sliven, Sliven
  - UHAT Aleksandrovska, Sofia
- North Macedonia (5):
  - PHI Clinical Hospital - Shtip, Department for Infectious Diseases and Febrile Conditions, Skopje
  - PHI General City Hospital "8mi Septemvri" - COVID-19 Intensive Care Department, Skopje
  - PHI University Clinic for Pulmonology and Allergology, Skopje
  - PHI University Clinic of Infectious Diseases and Febrile Conditions, Skopje
  - PHI General Hospital Struga bb, Quay "8-mi Noemvri", Struga
- University of Puerto Rico, San Juan, Puerto Rico
- South Korea (5):
  - Korea University Ansan Hospital, Ansan-si
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GLS-1027 120 mg | GLS-1027 360 mg | Placebo
Started | 42 | 46 | 44
Completed | 39 | 43 | 41
Not Completed | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GLS-1027 120 mg | GLS-1027 360 mg | Placebo | Total
Number analyzed (Participants) | 42 | 46 | 44 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 32 | 38 | 98
  >=65 years | 14 | 14 | 6 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (16.81) | 53.9 (15.38) | 52.2 (13.23) | 53.0 (15.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 27 | 82
  Male | 15 | 18 | 17 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 42 | 46 | 44 | 132
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 42 | 46 | 44 | 132
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  North Macedonia | 35 | 34 | 36 | 105
  Bulgaria | 7 | 11 | 7 | 25
  United States | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Events Relative to Treatment Group
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | GLS-1027 120 mg | GLS-1027 360 mg | Placebo
Number analyzed (Participants) | 42 | 46 | 44
participants | 1 | 3 | 0

2. Primary Outcome: Number of Treatment Failures at Day 28 From Enrollment
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | GLS-1027 120 mg | GLS-1027 360 mg | Placebo
Number analyzed (Participants) | 42 | 46 | 44
participants | 1 | 3 | 2

3. Secondary Outcome: Assess the Number of Days of Hospitalization Relative to Treatment Group
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | GLS-1027 120 mg | GLS-1027 360 mg | Placebo
Number analyzed (Participants) | 42 | 46 | 44
days | 9.3 (4.20) | 9.3 (3.65) | 9.4 (4.10)

4. Secondary Outcome: Assess the Number of Days Requiring ICU Care Relative to Treatment Group
Time Frame: 28 days
Measure: Mean (Inter-Quartile Range); unit: Days ICU care
Arm/Group | GLS-1027 120 mg | GLS-1027 360 mg | Placebo
Number analyzed (Participants) | 42 | 46 | 44
Days ICU care | 0 [0 to 0] | 4 [4 to 4] | 0 [0 to 0]

5. Secondary Outcome: Assess the Number of Days of NIV, High-flow O2, or Mechanical Ventilation Relative to Treatment Group
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | GLS-1027 120 mg | GLS-1027 360 mg | Placebo
Number analyzed (Participants) | 42 | 46 | 44
days | 6.7 (4.86) | 7.4 (4.43) | 6.1 (4.03)

6. Secondary Outcome: Assess the Maximal Level of Positive End-Expiratory Pressure (PEEP) for Subjects Who Are Intubated Relative to Treatment Group.
Time Frame: 28 days
Measure: Mean (Inter-Quartile Range); unit: cm H2O
Arm/Group | GLS-1027 120 mg | GLS-1027 360 mg | Placebo
Number analyzed (Participants) | 42 | 46 | 44
cm H2O | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

7. Secondary Outcome: Assess the Number of Days of PEEP > 5 cm H2O for Subjects Who Are Intubated Relative to Treatment Group
Time Frame: 28 days
Measure: Mean (Inter-Quartile Range); unit: Days intubated PEEP > 5 cm H2O
Arm/Group | GLS-1027 120 mg | GLS-1027 360 mg | Placebo
Number analyzed (Participants) | 42 | 46 | 44
Days intubated PEEP > 5 cm H2O | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent, daily while hospitalized (up to 15 days) and at days 28 and 56 by hospital records or telephone if discharged.
Arm/Group | GLS-1027 120 mg | GLS-1027 360 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/42 | 1/46 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/42 | 3/46 | 0/44
Other Adverse Events (participants affected / at risk) | 2/42 | 3/46 | 1/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLS-1027 120 mg (N=42) | GLS-1027 360 mg (N=46) | Placebo (N=44)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLS-1027 120 mg (N=42) | GLS-1027 360 mg (N=46) | Placebo (N=44)
Oral Candidiasis (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT04590547/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/47/NCT04590547/SAP_001.pdf